CLINICAL TRIAL: NCT01480050
Title: A Phase I Open Label Safety Study to Evaluate the Pharmacokinetic Profile and Tolerance of Mibefradil Dose Finding in Subjects With Recurrent High-Grade Glioma Undergoing Standard, Repeated Temozolomide Treatment
Brief Title: Mibefradil Dihydrochloride and Temozolomide in Treating Patients With Recurrent Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cavion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABTC-1101 CDR0000716313; NA_00068561 (Other: JHM IRB); M1 CA137443 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Brain Neoplasms | interventions — Temozolomide; alovudine; Mibefradil

ARMS (1):
- Dose Finding and Dose Expansion (Experimental): DOSE FINDING 4 Levels
  For all Levels:
  Cycle 1 Mibefradil QID dosing, Days 1-8 (to accommodate PKs) (*2 doses on Days 1 and 8) Temozolomide daily at 150-200 mg/m2, Days 9-13;
  Cycles 2+ Mibefradil QID, Days 1-7 Temozolomide daily at 150-200 mg/m2, Days 8-12
  DOSE EXPANSION 28-day cycles FLT PET scans, Baseline x2, Day 7 Mibefradil MTD determined at Dose Finding QID, Days 1-7 Temozolomide daily at 150-200 mg/m2, Days 8-12
  Interventions: Drug: temozolomide; Other: 3'-deoxy-3'-[18F]fluorothymidine; Other: pharmacological study; Drug: Mibefradil

INTERVENTIONS:
Drug: temozolomide — standard of care drug
Other: 3'-deoxy-3'-[18F]fluorothymidine — tracer used for FLT PET CT
Other: pharmacological study
Drug: Mibefradil

SUMMARY:
RATIONALE: Mibefradil dihydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the best dose of mibefradil dihydrochloride when given together with temozolomide in treating patients with glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum-tolerated dose (MTD) of mibefradil dihydrochloride administered prior to five days of temozolomide (TMZ) at 150-200 mg/m² in subjects with progressive or recurrent high-grade glioma.

Secondary

* Assess the safety of mibefradil dihydrochloride administered prior to five days of TMZ at 150-200 mg/m² when the mibefradil dihydrochloride dose is escalated from a starting dose of 100 mg/day, given four times a day for seven consecutive days.
* Determine the pharmacokinetic profile of mibefradil.
* Determine the steady state levels of mibefradil dihydrochloride on the last day of dosing.
* Assess the severity and frequency of adverse events for tested mibefradil dihydrochloride dose levels including cumulative toxicity and/or tolerance to adverse effects.
* Estimate the number and type of radiographic responses to treatment with mibefradil dihydrochloride and temozolomide.
* Assess the potential effect of mibefradil dihydrochloride on tumor metabolism as determined by Fluorothymidine Positron Emission Tomography (FLT PET) scans with the radiotracer [18F]-3'-fluoro-3'-deoxy-L-thymidine (dose-expansion cohort only).

OUTLINE: This is a dose-escalation study of mibefradil dihydrochloride followed by a dose-expansion study.

Patients receive mibefradil dihydrochloride orally (PO) 4 times a day on days 1-7 (days 1-8 on first course) and temozolomide PO on days 8-12 (days 9-13 on first course). Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected during the first course for pharmacokinetic studies.

Patients in the dose-expansion cohort undergo [18F]-3'-fluoro-3'-deoxy-L-thymidine (FLT)-positron emission tomography (PET) at baseline and on day 7 of the first course of therapy.

After completion of study therapy, patients are followed up every 2 months.

ELIGIBILITY:
ELIGIBILITY CRITERIA

* Subjects must be 18 years of age or older.
* Subjects must have histologically proven high-grade glioma (glioblastoma, anaplastic astrocytoma, anaplastic oligodendroglioma, mixed anaplastic oligoastrocytoma, anaplastic ependymoma) that is progressive or recurrent following standard upfront radiation therapy + temozolomide.
* Subjects must have measurable contrast-enhancing progressive or recurrent high grade glioma (single or multiple lesions) by MRI within 30 days of starting treatment.
* Subject must be able to tolerate MRIs. CT scans cannot be substituted for MRIs in this study.

  * Dose Expansion Subjects Only: the area of contrast enhancement must be at least 1 cm in short axis dimension.
* Subjects must have recovered to CTCAE grade <2 from toxicities related to prior therapy. An interval of at least 3 months must have elapsed since the completion of the most recent course of radiation therapy, the last dose of temozolomide (TMZ), or placement of Gliadel wafers. No prior cytotoxic therapies other than temozolomide and Gliadel wafers are allowed. Prior anti-VEGF therapies are allowed if more than four months have elapsed from the end of prior treatment. 30 days must have elapsed since previous treatment of the brain tumor with any other agents.
* Subjects must have a plan for retreatment with temozolomide at 150-200 mg/m2 for 5-days per cycle; each cycle = 28 days. Subjects must have previously tolerated at least one cycle of adjuvant temozolomide therapy in the prior treatment of the glioma (at 150-200 mg/m2 for 5 consecutive days).
* Subjects must have a Karnofsky Performance Status ≥ 60% (i.e. the subject must be able to care for himself/herself with occasional help from others).
* Subjects must have the following organ and marrow function:

  * Hemoglobin > 9 g/dL
  * Absolute neutrophil count >1,500/mcL
  * Platelets >100,000/mcL
  * Total bilirubin <3 times institutional upper limit of normal*
  * AST(SGOT)/ALT(SGPT) <3 times institutional upper limit of normal*
  * Creatinine within institutional upper limit of normal OR Creatinine clearance >50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
  * If above the institutional upper limit of normal but <3 times institutional upper limit of normal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient.
* Subjects must have serum potassium, magnesium, and calcium levels within normal institutional laboratory ranges (may be corrected to those levels by supplementation during screening period).
* Subjects must be able to provide written informed consent.
* Women of childbearing potential must have a negative pregnancy test prior to study entry. Women of childbearing potential and men must agree to use adequate contraception (adequate barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Subjects must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder.
* Subjects with prior malignancies must be disease-free for ≥ five years.
* Subjects must be maintained on a stable or decreasing corticosteroid regimen (no increase for 7 days) prior to the start of treatment.
* Subjects must identify a caregiver/support person who will agree to assist with the remote cardiac monitor and taking/recording blood pressure at home.

INELIGIBILITY CRITERIA

* Subjects with serious concurrent infection or medical illness, which would jeopardize the ability of the subject to receive the treatment outlined in this protocol with reasonable safety, are ineligible.
* Subjects may not be receiving any other investigational agents or chemotherapeutic agents other than temozolomide.
* Uncontrolled intercurrent illness including, but not limited to, hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women or those who are breastfeeding are ineligible.
* Subjects with a history of known, active hepatitis are ineligible.
* Subjects with a screening QTc interval greater than or equal to 450 mSec for males, 470 mSec for females are ineligible.
* Subjects with a PR interval >250 mSec are ineligible.
* Subjects with a systolic blood pressure <100 mmHg at baseline are ineligible.
* Subjects taking any anti-arrhythmia medication other than beta-blockers or digoxin or with a history (within six months) of myocardial infarction, unstable angina, uncontrolled hypertension, or congestive heart failure are ineligible.
* Subjects with high grade (second degree or above) AV block or persistent sinus bradycardia of less than 50 BPM are ineligible.
* Subjects who require a calcium channel blocker for blood pressure control and who cannot be switched to an antihypertensive with an alternative mechanism of action will be excluded from the study. Permitted anti-hypertensive medications include:

  * chlorothiazide
  * hydrochlorothiazide
  * atenolol
  * nadolol
  * enalapril
  * lisinopril,
  * eprosartan
  * irbesartan.
* Subjects cannot receive any statin while on trial except pravastatin.
* Subjects who require treatment with an H2 blocker, other than famotidine, are ineligible. If the subject requires a proton pump inhibitor (PPI), then esomeprazole, pantoprazole, or rabeprazole may be given.
* Known HIV-positive subjects are ineligible because of potential CNS conditions associated with HIV and the possibility of unexpected drug-drug interactions.
* Subjects on enzyme-inducing anti-epileptic drugs (EIAEDs) are not eligible for treatment on this protocol. Subjects previously treated with EIAEDs may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of mibefradil.
* Subjects taking an anticoagulant must use warfarin or a low molecular weight heparin. Unfractionated heparin is not permitted. Appropriate monitoring of the effect of anticoagulation is required by guidelines.
* All subjects who require drugs that are substrates of CYP 3A4, CYP 2D6, and CYP 1A2 are ineligible except for the ones that are explicitly permitted
* Subjects who require any drugs that are known to interact adversely with metabolism or excretion of mibefradil are ineligible.
* Subjects who are taking and cannot discontinue over-the-counter (OTC) medications and nutritional supplements, including herbal or "Chinese" medications are ineligible.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of mibefradil dihydrochloride | 2 years
  Determine the maximum tolerated dose (MTD) of mibefradil administered prior to five days of temozolomide (TMZ) at 150-200 mg/m2 in subjects with progressive or recurrent high grade glioma.
Dose-limiting toxicity | 2 years

SECONDARY OUTCOMES:
Toxicity and adverse events according to CTCAE v. 4.0 | 2 years
  Assess the severity and frequency of adverse events for tested mibefradil dose levels including cumulative toxicity and/or tolerance to adverse effects.
Biological activity of treatment determined by radiographic response | 3 years
  Estimate the number and type of radiographic responses to treatment with mibefradil and temozolomide.
Pharmacokinetics of mibefradil dihydrochloride as measured by the steady-state maximum plasma concentration (Cmax) | Day 8
  Cmax (ng/mL) of mibefradil dihydrochloride at steady-state in plasma.
Potential effect of mibefradil dihydrochloride on tumor metabolism as determined by [F-18]FLT PET scans in the dose-expansion cohort | 6 months
  Assess the potential effect of mibefradil on tumor metabolism as determined by fluorothymidine positron emission tomography-computed tomography (FLT PETCT) scans with the radiotracer [18F]-3'-fluoro-3'-deoxy-L-thymidine.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Holdhoff, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (7):
- United States (7):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Holdhoff M, Ye X, Supko JG, Nabors LB, Desai AS, Walbert T, Lesser GJ, Read WL, Lieberman FS, Lodge MA, Leal J, Fisher JD, Desideri S, Grossman SA, Wahl RL, Schiff D. Timed sequential therapy of the selective T-type calcium channel blocker mibefradil and temozolomide in patients with recurrent high-grade gliomas. Neuro Oncol. 2017 Jun 1;19(6):845-852. doi: 10.1093/neuonc/nox020. PMID 28371832